CLINICAL TRIAL: NCT01811277
Title: Phase II Exploratory Study of S-1 Combined With Oxaliplatin Sequential S-1 Single-agent First-line Treatment of Unresectable Metastatic or Locally Advanced Biliary System, Periampullary Cancer and Pancreatic Cancer
Brief Title: SOX Sequential S-1 in Advanced Biliary Tract Carcinoma（BTC）and Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Head of GI Cancer department, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOX-S-1 BTC
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2010-07

CONDITIONS: Biliary Tract Cancer; Periampullary Adenocarcinoma; Pancreatic Cancer
Keywords: palliative chemotherapy; ORR; PFS; OS; safety; advanced Biliary Tract Carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOX sequential S-1 (Experimental): 4-6 cycles of SOX followed by S-1 monotherapy until disease progression
  Interventions: Drug: SOX sequential S-1

INTERVENTIONS:
Drug: SOX sequential S-1 — 4-6 cycles SOX followed by S-1 monotherapy until disease progression
  S-1: 40~60mg bid，po, d1~14 （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid） oxaliplatin：130mg/m2，iv drip for 2h，d1
  Other Names: S-1/oxaliplatin

SUMMARY:
This is an exploratory, single-armed, open label study on the efficacy and safety of sequential S-1 therapy after SOX in unresectable metastatic or locally advanced biliary system or periampullary cancer or pancreatic cancer patients. The primary endpoint is Objective response rate and secondary endpoint is progression free survival , overall survival ,1 year survival rate and safety.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Male or female patients >=18 years old
* Histologically or cytologically confirmed diagnosis of adenocarcinoma
* No previous treatment is allowed including chemotherapy, radiotherapy,immunotherapy or others.
* In case the patient received adjuvant therapy before, enrollment is allowed if the adjuvant therapy does not contain L-OHP or S-1 and at the same time, the last day of chemotherapy is ≥180 days before screening.
* Target lesion more than 1cm in diameter by enhanced CT or MRI 21 days before enrollment
* The laboratory parameter meets the following criteria 7 days before enrollment

  * Hemoglobin ≥90g/L
  * Absolute neutrophil count≥1.5×10^9/L, platelets 100×10^9/L；
  * ALT and AST≤2.5 ULN(in case of the patients with liver metastasis,ALT and AST≤5.0 ULN)
  * ALP ≤2.5 ULN (in case of the patients with liver metastasis,≤5.0 ULN)
  * Total Serum bilirubin ≤1.5 ULN
  * Serum creatinine ≤1.0 ULN
  * serum albumin(ALB)≥30g/L；
* can tolerate oral drug administration；
* KPS ≥70
* Estimated survival ≥90 days
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of enrollment and must be willing to use adequate methods of contraception during the study and for 30 days after last study durg administration.

Exclusion Criteria:

* Known sensitivity to 5-HT3 antagonist and hypersensitivity to the other treatment agents including irinotecan, cisplatin and octreotide lar
* Any participation in trials simultaneously or 4 weeks before screening.
* 15 days prior to enrollment, received a blood transfusion, blood products and hematopoietic growth factors such as G-CSF.
* Undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such surgery.
* Uncontrolled severe diarrhea
* Uncontrolled active infection (fever ≥38 degrees due to infection)
* S-1 oral drug administration difficulty due to difficulty swallowing, complete or incomplete digestive tract obstruction, gastrointestinal active bleeding, perforation;
* severe hepatopathy including active hepatitis and hepatic cirrhosis, renal dysfunction, severe pulmonary diseases including interstitial pneumonia, pulmonary fibrosis and severe pulmonary emphysema, uncontrolled diabetes, hypertension and other chronic systematic diseases.
* Chronic treatment with steroids.(In case of the patients with short-term use of steroids, the enrollment is permitted if the administration is stopped 2 weeks before screening.)
* confirmed or suspected CNS metastasis
* the history of peripheral nervous system impairment, obvious mental disorder or CNS impairment
* clinically significant heart disease, including congestive heart failure, symptomatic coronal heart disease, arrythmia uncontrolled by medication and acute myocardial infarction or cardiac insufficiency within 6 months before screening
* Drainage of pleural effusion, peritoneal effusion and pericardial effusion
* pregnant women or women in lactation period
* Fertile male or women of child-bearing potential refuse to take highly effective methods of birth control
* Incidence of other second primary malignant tumors within 5 years, except for cured basal cell carcinoma and cervical carcinoma in situ.
* patients of legal incapacity or who have the potential of influence the whole trial due to medical or ethic reasons.
* Other patients who are not eligible to the trial under investigators' discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate for SOX sequential S-1 | 1 years
  The primary endpoint is objective response rate,which equals CR+PR.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost
progression free survival | 1 year
  PFS means that from the first dose of treatment drug to disease progression or death or lost, the follow-up visit will be performed every 6 weeks till progression or death or lost
1 year survival rate | 1 year
  the follow-up visit of survival will be performed every 3 months till 1 year
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
  participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Prof., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China